CLINICAL TRIAL: NCT05578339
Title: Predicting the Lens Capsular Bag Size Using Pre-operative Biometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, head of department of Ophthalmology, Professor, Principal Investigator, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Capsular bag size
Record Dates: First submitted 2022-01-30; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Cataract Senile
Keywords: capsular bag
MeSH Terms: interventions — Biometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capsular bag size (Other): Lens thickness, lens shape, anterior chamber depth, axial eye length and angle-to-angle will be used as explanatory variables (independent variables) and the size of the capsular bag will be used as main outcome parameter (dependent variable).
  We will perform a multiple linear regression analysis (that allows determination of the overall fit (variance explained) of the model and the relative contribution of each of the predictors to the total variance explaine) between the independent and the dependent variable.
  Interventions: Device: Biometry

INTERVENTIONS:
Device: Biometry — Lens thickness, lens shape, anterior chamber depth, axial eye length and angle-to-angle will be used as explanatory variables (independent variables) and the size of the capsular bag will be used as main outcome parameter (dependent variable).

SUMMARY:
Aim of this study is to assess whether a high-resolution scan of the crystalline lens before surgery may be helpful in predicting post-operative capsule bag diameter.

DETAILED DESCRIPTION:
Most of the measurement procedures used in this study are non-invasive and all are used in standard routine clinical practice, the benefit/risk ratio appears acceptable.

However, a capsule tension ring will be used. A CTR is not used routinely, usually only in cataract operations in which the lens capsule is not stable enough - in other words, for stabilization. The insertion of the CTR is problem-free in most cases. In extremely rare cases, however, the lens capsule may be injured. And document complications will be collected, report them in a final paper. The CTR used in the study is a standard device and CE-marked device. Studies using CTR showed that it is beneficial in difficult cases.

Gonioscopy after cataract surgery will be performed after 1 week. At this time point the wound is already sealed and there appears to be no increased risk to the patient. In the first study performed in a similar fashion in 1999 gonioscopy was performed one day after surgery.

Aim of this study is to predict the diameter of the capsular bag using pre-operative optical biometry findings.

This is a prospective, observer-blind and monocentric study that includes patients scheduled for cataract surgery. Recruitment will take part on the day of pre-assessment. For each patient only one eye will be included.

In total 50 eyes of 50 patients will be included, of which at least 5 eyes with an axial eye length below 22.5mm and 5 eyes with an axial eye length above 25.0mm.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for cataract surgery
* Well dilated pupil at the pre-assessment visit (dilated pupil size at least 6.0mm)
* Age 21 and older
* Pre-operative visual acuity of at least 0.25 Snellen

Exclusion Criteria:

* Parameters that influence the capsular bag stability (pseudoexfoliation syndrome, St. p. severe eye trauma, Phakodonesis)
* In women of childbearing age, a pregnancy test will be performed before inclusion into the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Capsular bag size | 2 months
  • Prediction of the size of the post-operative capsular bag diameter using pre-operative optical biometry (lens thickness, lens shape, anterior chamber depth, axial eye length and angle-to-angle distance)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
all results will be published